CLINICAL TRIAL: NCT04237298
Title: Comparison of Relapse Arch Width in Modified Vacuum Formed Retainers Covering the Palate Versus Hawley Retainer: A Prospective Randomized Control Trial
Brief Title: Comparison of Modified Vacuum-formed Retainers Versus Hawley Retainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, ASMA ASHARI, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GGPM-2018-049
Record Dates: First submitted 2019-10-04; First posted 2020-01-23 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Orthodontic Retainers; Clinical Trial
Keywords: Space Maintenance; Palatal Expansion Technique; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hawley retainer (Active Comparator): Standard retention regime for patients with arch expansion. Patients will be instructed to wear the retainer 24 hours during the study period.
  Interventions: Device: Modified vacuum-formed retainer covering the palete
- Modified vacuum-formed retainer covering the palate (Experimental): The modified vacuum-formed retainer is designed to cover the palate. It is cheaper, easier to fabricate and more esthetic. Patients will be instructed to wear the retainer 24 hours during the study period.
  Interventions: Device: Modified vacuum-formed retainer covering the palete

INTERVENTIONS:
Device: Modified vacuum-formed retainer covering the palete — The modified vacuum-formed retainer is made where it would cover the hard palate to the second molars. The only difference in constructing this modified VFR when compared to the normal VFR would be the outline which would be trimmed by the technician.
  Other Names: Essix retainer covering the palate; Thermoplastic retainer covering the palate

SUMMARY:
This study will focus on the relapse of arch width in two types of retention regimes, which are modified vacuum-formed retainers and Hawley type retainers in patients after fixed appliance treatment in transverse arch expansion cases. This will subsequently be of valuable information for clinicians in choosing the appropriate type of retainers after removal of their fixed appliances. This is because the modified vacuum-formed retainers will be significantly cheaper, quicker and easier to fabricate.

DETAILED DESCRIPTION:
Relapse is inevitable in orthodontic treatment. Teeth will want to return to their original position after fixed appliances are removed. Regardless with or without fixed appliances, changes and physiological relapse will still occur due to time and age changes. This is why retention is a crucial part of orthodontic treatment, where it would aim to maintain the corrections achieved after orthodontic treatment.

Literature regarding retainers is quite substantial, where a recent Cochrane review was published comparing the different types of retainers. However, the evidence is lacking in terms of comparison of arch width relapse between modified vacuum-formed retainers and Hawley retainers specifically in expansion cases.

This study aims to compare the relapse in arch width in expansion cases with modified vacuum-formed retainers with palatal coverage versus Hawley type retainers in Unit Ortodontik Universiti Kebangsaan Malaysia (UKM), Klinik Pakar Ortodontik Klinik Kesihatan Bandar Botanik and Unit Pakar Ortodontik Klinik Pergigian Sungai Chua patients. Although other types of modified vacuum-formed retainers effective for maintaining palatal expansion have been described, these retainers require a wire outlining the Cementoenamel junction of the teeth palatally. This technique requires the experience of the technician, is at a higher cost and requires more lab time. The modified retainer that investigators described in this study would be as efficient and as quick as the normal vacuum-formed retainers, which would usually take a couple of hours to make (same day or next day fit). The present practice at all 3 locations constructs Hawley and normal VFR retainers for all orthodontic patients. There are technicians and laboratory facilities to construct normal VFR as well as Hawley retainer. The only difference between modified and normal vacuum formed retainer is the outline of the retainers where the technician would trim the retainer, where it would cover the hard palate. Therefore it is only the location of trimming that is different using the same special trimming appliances for normal VFRs.

A number of subjects who fulfil the criteria will be invited to participate in this study. The study will involve arch width analysis using study models pre, post-debond, 3 months review post-debond, and 6 months review post-debond. All data will be analyses using Statistical Package for Social Sciences (SPSS). The arch width of participants post-fixed appliances will be compared. Most studies compare the arch width, as well as lower incisor irregularity in evaluating relapse in different groups of retainers. However, there are currently no randomized control trials comparing expansion cases of Hawley vs vacuum-formed retainers, hence why this study will be conducted.

The investigators expect to see no difference between the modified vacuum formed retainer and Hawley retainer in terms of maintaining arch expansion post-orthodontic treatment. This would, therefore, mean that there would be a simpler method and would be a suitable more cost-effective alternative as compared to constructing Hawley retainers or adding a palatal wire on the vacuum-formed retainers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are at least 13 years old at time of debond.
2. Treatment plan of extraction or non-extraction followed by straight wire appliances in the upper arch only or both arches
3. Undergone more than 3mm of maxillary dentoalveolar expansion. Initially, the amount of arch width expansion was measured intraorally at debond and compared to their respective pre-treatment dental casts. To ensure accuracy, the measurements were repeated on debond and pre-treatment dental casts. The following linear arch width measurements were made: intercanine width (ICW - the distance between the canine cusp tips), interpremolar width (IPMW - the distance between the premolar cusp tips), interfirst molar width 1 (IFMW1 - the distance between the mesiobuccal cusp), and interfirst molar width 2 (IFMW2 - the distance between the distobuccal cusp). At least two or more points were expanded (> 3mm) to be included in the trial.
4. No chronic medical conditions

Exclusion Criteria:

-

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DR. ASMA ASHARI, Principal Investigator — National University of Malaysia
Locations (3):
- Malaysia (3):
  - Unit Pakar Ortodontik Klinik Pergigian Sungai Chua, Kajang, Selangor
  - Klinik Pakar Ortodontik Klinik Kesihatan Bandar Botanik, Klang, Selangor
  - Orthodontic Specialist Clinic, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment : 1 Aug 2019 til 31st Aug 221
Pre-assignment Details: Excluded: not meeting inclusion criteria, declined to participate
Groups:
- Hawley Retainer: Standard retention regime for patients with arch expansion. Patients will be instructed to wear the retainer 24 hours during the study period.
  Hawley retainer: Standard retention regime for patients with arch expansion. Patients will be instructed to wear the retainer 24 hours during the study period.
Period: Overall Study
Arm/Group | Hawley Retainer | Modified Vacuum-formed Retainer Covering the Palate
Started | 17 | 18
Completed | 13 | 13
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hawley Retainer | Modified Vacuum-formed Retainer Covering the Palate | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.88 (4.12) | 22.06 (5.88) | 21.97 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Arch Width
Description: Mean changes across 24-month study period.
Time Frame: 24-month post-debond
Population: arch width (transverse)
Measure: Mean (95% Confidence Interval); unit: milimeters
Arm/Group | Hawley Retainer | Modified Vacuum-formed Retainer Covering the Palate
Number analyzed (Participants) | 17 | 18
milimeters
  intercanine width | 36.9 [35.76 to 38.04] | 37.65 [36.54 to 38.76]
  interpremolar width | 44.61 [43.39 to 45.82] | 46.31 [45.09 to 47.52]
  interfirst molar width 1 | 50.74 [49.64 to 51.85] | 52.86 [51.82 to 53.90]
  interfirst molar width 2 | 52.04 [50.78 to 53.31] | 54.05 [52.86 to 55.25]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse event was not monitored
Arm/Group | Hawley Retainer | Modified Vacuum-formed Retainer Covering the Palate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04237298/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04237298/ICF_001.pdf